CLINICAL TRIAL: NCT02993822
Title: A Double-Blind, Randomized, Placebo Controlled Study of the Efficacy and Safety of Three Doses of Orvepitant in Subjects With Chronic Refractory Cough
Brief Title: A Dose-ranging Study of Orvepitant in Patients With Chronic Refractory Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nerre Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VOLCANO-2
Record Dates: First submitted 2016-12-06; First posted 2016-12-15 (Estimated); Results first posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-03

CONDITIONS: Chronic Refractory Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orvepitant 10mg (Experimental): Orvepitant 10mg tablet, once daily for 12 weeks
  Interventions: Drug: Orvepitant Maleate
- Orvepitant 20mg (Experimental): Orvepitant 20mg tablet, once daily for 12 weeks
  Interventions: Drug: Orvepitant Maleate
- Orvepitant 30mg (Experimental): Orvepitant 30mg tablet, once daily for 12 weeks
  Interventions: Drug: Orvepitant Maleate
- Placebo (Placebo Comparator): Placebo to match tablet, once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orvepitant Maleate — Tablet, once daily, oral
  Arms: Orvepitant 10mg; Orvepitant 20mg; Orvepitant 30mg
Drug: Placebo — Tablet, once daily, oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of three doses of orvepitant, taken once a day, in the treatment of chronic refractory cough.

DETAILED DESCRIPTION:
A multi-center, double-blind, randomized, parallel group, placebo-controlled dose range study in subjects with chronic refractory cough (CRC).

Doses of orvepitant (10 mg/day, 20 mg/day and 30 mg/day) and placebo will be investigated in four parallel groups.

Each group will compromise of approximately 73 subjects, randomized 1:1:1:1 (approximately 292 subjects in total).

All subjects will enter a three-week screening period to determine eligibility. Eligible subjects will be randomized at the Baseline/Day 1 visit and enter a 12-week double-blind dosing period. During this period there will be four visits at Weeks 2, 4, 8 and 12. There will be a final safety follow-up visit at Week 14.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female subjects ≥18 years of age.
* Diagnosis of CRC or unexplained cough for at least 1 year (see ACCP/BTS guidelines attached).
* An awake average cough frequency of ≥10 coughs/ hour, as assessed using an ACM during the screening period.

Key Exclusion Criteria:

* Subjects with respiratory tract infection (<4 weeks prior to study start)
* Current smokers or ex-smokers with <6 months' abstinence or cumulative history of >10 pack years
* Treatment with Angiotensin Converting Enzyme (ACE) inhibitors within 3 months of screening
* FEV1 <80% predicted, measured at screening using spirometry
* History of cystic fibrosis, idiopathic pulmonary fibrosis, clinically significant bronchiectasis, moderate to severe asthma, chronic obstructive pulmonary disease (COPD)
* Any clinically significant abnormal laboratory test result(s)
* Inability to comply with the use of prohibited and allowed medications as described in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (46):
  - Study Site 15, Chandler, Arizona
  - Study Site 43, Los Angeles, California
  - Study Site 52, Mission Viejo, California
  - Study Site 20, San Diego, California
  - Study Site 28, San Jose, California
  - Study Site 25, Centennial, Colorado
  - Study Site 36, Colorado Springs, Colorado
  - Study Site 48, Waterbury, Connecticut
  - Study Site 68, Clearwater, Florida
  - Study Site 59, Jacksonville, Florida
  - Study Site 12, Largo, Florida
  - Study Site 62, Miami, Florida
  - Study Site 57, Miami, Florida
  - Study Site 33, Tampa, Florida
  - Study Site 11, Winter Park, Florida
  - Study Site 60, Meridian, Idaho
  - Study Site 39, Normal, Illinois
  - Study Site 34, Baltimore, Maryland
  - Study Site 42, Edina, Minnesota
  - Study Site 41, Minneapolis, Minnesota
  - Study Site 37, Rochester, Minnesota
  - Study Site 27, Missoula, Montana
  - Study Site 16, Las Vegas, Nevada
  - Study Site 32, Rochester, New York
  - Study Site 55, Charlotte, North Carolina
  - Study Site 24, Charlotte, North Carolina
  - Study Site 53, Charlotte, North Carolina
  - Study Site 50, Gastonia, North Carolina
  - Study Site 54, Greensboro, North Carolina
  - Study Site 73, Mooresville, North Carolina
  - Study Site 71, Raleigh, North Carolina
  - Study Site 56, Cincinnati, Ohio
  - Study Site 74, Oklahoma City, Oklahoma
  - Study Site 26, Tulsa, Oklahoma
  - Study Site 38, East Providence, Rhode Island
  - Study Site 21, Charleston, South Carolina
  - Study Site 72, Charleston, South Carolina
  - Study Site 22, Dallas, Texas
  - Study Site 35, Dallas, Texas
  - Study Site 10, Houston, Texas
  - Study Site 49, San Antonio, Texas
  - Study Site 23, Waco, Texas
  - Study Site 58, Salt Lake City, Utah
  - Study Site 19, Charlottesville, Virginia
  - Study Site 14, Bellingham, Washington
  - Study Site 13, Greenfield, Wisconsin
- Canada (3):
  - Study Site 66, Niagara Falls, Ontario
  - Study Site 65, Québec, Quebec
  - Study Site 64, Trois-Rivières, Quebec
- United Kingdom (17):
  - Study Site 29, Romford, Essex
  - Study Site 94, Blackpool, Lancashire
  - Study Site 93, Prescot, Merseyside
  - Study Site 17, Northwood, Middlesex
  - Study Site 40, Belfast, Northern Ireland
  - Study Site 96, Barnsley, South Yorkshire
  - Study Site 97, Cannock, Staffordshire
  - Study Site 95, Stockton-on-Tees, Teesside
  - Study Site 45, Hull
  - Study Site 92, Leeds
  - Study Site 30, Leicester
  - Study Site 46, London
  - Study Site 91, Manchester
  - Study Site 18, Manchester
  - Study Site 47, Newcastle upon Tyne
  - Study Site 31, North Shields
  - Study Site44, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled (screened and consented) on 22-May-2017; the first subject was randomised on 31-Jan-2017. The last subject was enrolled on 28-Sep-2018. The last subject last visit (study completion) was 24-Jan-2019.
  Subjects were recruited from a mixture of specialised standalone clinics and clinics within hospitals.
Pre-assignment Details: Screening details:
  488 subjects were screened, of whom 315 (64.5%) completed screening and were randomised.
  Screening failures occurred due to not meeting inclusion criteria (74 subjects [15.2%]) or exclusion criteria (79 subjects [16.2%]), withdrawal of consent (nine [1.8%] subjects) and AEs (2 [0.4%] subjects). All other reasons reported in individual subjects.
Period: Overall Study
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Started | 79 | 78 | 79 | 79
Completed | 69 | 74 | 69 | 75
Not Completed | 10 | 4 | 10 | 4
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Unable to attend follow-up due to illness | 0 | 0 | 0 | 1
Not completed — Adverse Event | 3 | 1 | 7 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 2 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo | Total
Number analyzed (Participants) | 79 | 78 | 79 | 79 | 315
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 44 | 56 | 37 | 183
  >=65 years | 33 | 34 | 23 | 42 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.29 (9.850) | 59.86 (13.173) | 59.47 (10.020) | 62.24 (11.815) | 60.97 (11.313)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 69 | 60 | 59 | 253
  Male | 14 | 9 | 19 | 20 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 4 | 6
  Not Hispanic or Latino | 74 | 74 | 77 | 74 | 299
  Unknown or Not Reported | 5 | 3 | 1 | 1 | 10
Region of Enrollment [Number; unit: participants]
  North America | 51 | 49 | 51 | 51 | 202
  Europe | 28 | 29 | 28 | 28 | 113

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Awake Objective Cough Frequency
Description: Objective cough frequency measured by ambulatory cough monitoring device
Time Frame: Baseline to Week 12
Population: The number of participants analyzed differs from the overall subject disposition as it includes only participants with data available for the comparison (i.e. some participants have missing data).
Measure: Mean (Standard Deviation); unit: coughs per hour (log transformed)
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 66 | 72 | 67 | 70
coughs per hour (log transformed) | -0.185 (0.3258) | -0.192 (0.3405) | -0.271 (0.4055) | -0.243 (0.3225)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; Change from baseline to each visit (Week 2, Week 4 and Week 12) in log transformed awake objective cough frequency was analysed using a mixed model for repeated measures (MMRM) with restricted maximum likelihood (REML) estimation. The treatment effect at Week 12 was estimated using the ratio of geometric means (i.e. the difference between the treatments least squares means [adjusted means] on the log scale, back transformed to the original scale); Test type: Superiority; p = 0.324, Mixed model repeated measures; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [0.88 to 1.49]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.332, Mixed model repeated measures; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [0.88 to 1.48]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.531, Mixed model repeated measures; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [0.71 to 1.20]

2. Secondary Outcome: Change in Awake Objective Cough Frequency at Week 2 Compared to Baseline
Description: Objective cough frequency measured by ambulatory cough monitoring device
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: coughs per hour (log transformed)
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 73 | 74 | 75 | 73
coughs per hour (log transformed) | -0.180 (0.2791) | -0.181 (0.3142) | -0.215 (0.2515) | -0.139 (0.2892)
Statistical Analysis 1: Comparison: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.482, Mixed model repeated measures; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [0.75 to 1.15]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.460, Mixed model repeated measures; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [0.75 to 1.14]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.144, Mixed model repeated measures; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [0.69 to 1.06]

3. Secondary Outcome: Change in Awake Objective Cough Frequency at Week 4 Compared to Baseline
Description: Objective cough frequency measured by ambulatory cough monitoring device
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: coughs per hour (log transformed)
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 68 | 77 | 75 | 72
coughs per hour (log transformed) | -0.188 (0.3292) | -0.231 (0.3665) | -0.211 (0.2994) | -0.169 (0.2699)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.992, Mixed model repeated measures; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [0.78 to 1.27]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.387, Mixed model repeated measures; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [0.71 to 1.14]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.600, Mixed model repeated measures; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [0.74 to 1.19]

4. Secondary Outcome: Change in the Leicester Cough Questionnaire (LCQ) at Week 2 Compared to Baseline
Description: The Leicester Cough Questionnaire (LCQ) is a 19 item questionnaire that assessed cough related quality of life. It has three domains (physical, psychological and social) and subjects were asked to complete it based on their experience in a recall period of 2 weeks. The total score range is 3 to 21 and domain scores each range from 1 to 7; a higher score indicated a better quality of life. Subjects completed the LCQ whilst in the clinic at baseline/Day 1 (pre dose) and at Weeks 2, 4, 8, and 12.
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 72 | 77 | 75 | 75
Total score | 2.41 (3.309) | 2.37 (3.252) | 2.93 (3.010) | 1.24 (2.714)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; The change from baseline in LCQ total score and the three domain scores was summarised by treatment group and visit (Weeks 2, 4, 8 and 12) in terms of absolute values and changes from baseline. The effect of treatment in terms of the change from baseline to each scheduled visit (Week 2, Week 4, Week 8 and Week 12) in LCQ total score and the three domain scores was analysed using a MMRM with REML estimation; Test type: Superiority; p = 0.042, Mixed model repeated measures; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.0 to 2.0]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.026, Mixed model repeated measures; Median Difference (Final Values) = 1.1, 95% CI 2-sided [0.1 to 2.0]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.003, Mixed model repeated measures; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [0.5 to 2.4]

5. Secondary Outcome: Change in the Leicester Cough Questionnaire (LCQ) at Week 4 Compared to Baseline
Description: The Leicester Cough Questionnaire (LCQ) is a 19 item questionnaire that assessed cough related quality of life. It has three domains (physical, psychological and social) and subjects were asked to complete it based on their experience in a recall period of 4 weeks. The total score range is 3 to 21 and domain scores each range from 1 to 7; a higher score indicated a better quality of life. Subjects completed the LCQ whilst in the clinic at baseline/Day 1 (pre dose) and at Weeks 2, 4, 8, and 12.
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 68 | 77 | 74 | 76
Total score | 2.50 (3.416) | 2.15 (3.490) | 2.98 (3.163) | 1.61 (3.132)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.250, Mixed model repeated measures; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.4 to 1.7]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.325, Mixed model repeated measures; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.5 to 1.5]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.029, Mixed model repeated measures; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [0.1 to 2.2]

6. Secondary Outcome: Change in the Leicester Cough Questionnaire (LCQ) at Week 8 Compared to Baseline
Description: The Leicester Cough Questionnaire (LCQ) is a 19 item questionnaire that assessed cough related quality of life. It has three domains (physical, psychological and social) and subjects were asked to complete it based on their experience in a recall period of 8 weeks. The total score range is 3 to 21 and domain scores each range from 1 to 7; a higher score indicated a better quality of life. Subjects completed the LCQ whilst in the clinic at baseline/Day 1 (pre dose) and at Weeks 2, 4, 8, and 12.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 66 | 76 | 70 | 75
Total score | 2.78 (3.535) | 2.19 (3.602) | 2.82 (3.960) | 1.34 (3.222)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.038, Mixed model repeated measures; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.1 to 2.3]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.118, Mixed model repeated measures; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.2 to 2.0]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.025, Mixed model repeated measures; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.2 to 2.4]

7. Secondary Outcome: Change in the Leicester Cough Questionnaire (LCQ) at Week 12 Compared to Baseline
Description: The Leicester Cough Questionnaire (LCQ) is a 19 item questionnaire that assessed cough related quality of life. It has three domains (physical, psychological and social) and subjects were asked to complete it based on their experience in a recall period of 12 weeks. The total score range is 3 to 21 and domain scores each range from 1 to 7; a higher score indicated a better quality of life. Subjects completed the LCQ whilst in the clinic at baseline/Day 1 (pre dose) and at Weeks 2, 4, 8, and 12.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 66 | 74 | 67 | 74
Total score | 2.38 (3.609) | 2.09 (3.736) | 3.23 (4.007) | 1.50 (3.586)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.258, Mixed model repeated measures; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.5 to 1.9]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.243, Mixed model repeated measures; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.5 to 1.8]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.009, Mixed model repeated measures; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [0.4 to 2.8]

8. Secondary Outcome: Change in the Cough Severity Visual Analogue Scale (VAS) at Week 2 Compared to Baseline - Day-time
Description: The cough VAS is a 100 mm scale on which subjects indicated their severity of cough over the previous 24 hours, both during the day-time and during night time separately. The VAS ranged from "no cough" (0 mm) on the left to "worst cough" (100 mm) on the right. Subjects completed the cough severity VAS at baseline/Day 1 (pre dose) and at Weeks 2, 4, 8, and 12.
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 71 | 77 | 75 | 75
Score | -17.7 (26.06) | -10.5 (27.78) | -13.5 (22.93) | -6.3 (19.24)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; Change in the Cough Severity VAS was summarised by treatment group and visit (Weeks 2, 4, 8 and 12) in terms of absolute values and changes from baseline. The effect of treatment in terms of the change from baseline to each scheduled visit (Week 2, Week 4, Week 8 and Week 12) in Cough Severity VAS was analysed using a MMRM with REML estimation; Test type: Superiority; p = 0.008, Mixed model repeated measures; Mean Difference (Final Values) = -9.6, 95% CI 2-sided [-16.6 to -2.5]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.198, Mixed model repeated measures; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-11.4 to 2.4]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.055, Mixed model repeated measures; Mean Difference (Final Values) = -6.8, 95% CI 2-sided [-13.7 to 0.1]

9. Secondary Outcome: Change in the Cough Severity Visual Analogue Scale (VAS) at Week 4 Compared to Baseline - Day-time
Description: as for outcome 8
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 68 | 77 | 75 | 76
Score | -17.9 (27.11) | -9.4 (26.76) | -15.9 (25.02) | -7.8 (22.36)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.026, Mixed model repeated measures; Mean Difference (Final Values) = -8.7, 95% CI 2-sided [-16.3 to -1.1]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.571, Mixed model repeated measures; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-9.6 to 5.3]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.043, Mixed model repeated measures; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-15.2 to -0.3]

10. Secondary Outcome: Change in the Cough Severity Visual Analogue Scale (VAS) at Week 8 Compared to Baseline - Day-time
Description: as for outcome 8
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 66 | 76 | 72 | 75
Score | -21.0 (30.37) | -9.9 (29.57) | -18.6 (27.24) | -8.2 (23.58)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.006, Mixed model repeated measures; Mean Difference (Final Values) = -11.5, 95% CI 2-sided [-19.7 to -3.3]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.435, Mixed model repeated measures; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-11.1 to 4.8]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.022, Mixed model repeated measures; Mean Difference (Final Values) = -9.4, 95% CI 2-sided [-17.4 to -1.4]

11. Secondary Outcome: Change in the Cough Severity Visual Analogue Scale (VAS) at Week 12 Compared to Baseline - Day-time
Description: as for outcome 8
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 66 | 74 | 68 | 73
Score | -18.8 (31.27) | -11.6 (27.33) | -20.1 (29.33) | -10.6 (24.46)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.103, Mixed model repeated measures; Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-15.3 to 1.4]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.546, Mixed model repeated measures; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-10.6 to 5.6]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.034, Mixed model repeated measures; Mean Difference (Final Values) = -9.0, 95% CI 2-sided [-17.2 to -0.7]

12. Secondary Outcome: Change in the Cough Severity Visual Analogue Scale (VAS) at Week 2 Compared to Baseline - Night-time
Description: as for outcome 8
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 71 | 77 | 75 | 75
Score | -12.8 (28.96) | -7.8 (26.76) | -6.2 (24.97) | -3.9 (27.62)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.004, Mixed model repeated measures; Mean Difference (Final Values) = -11.2, 95% CI 2-sided [-18.8 to -3.6]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.282, Mixed model repeated measures; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-11.5 to 3.4]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.398, Mixed model repeated measures; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-10.7 to 4.3]

13. Secondary Outcome: Change in the Cough Severity Visual Analogue Scale (VAS) at Week 4 Compared to Baseline - Night-time
Description: as for outcome 8
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 68 | 77 | 75 | 76
Score | -10.1 (32.87) | -7.9 (27.52) | -5.8 (27.96) | -2.7 (27.99)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.019, Mixed model repeated measures; Mean Difference (Final Values) = -10.0, 95% CI 2-sided [-18.3 to -1.7]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.170, Mixed model repeated measures; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-13.7 to 2.4]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.384, Mixed model repeated measures; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-11.7 to 4.5]

14. Secondary Outcome: Change in the Cough Severity Visual Analogue Scale (VAS) at Week 8 Compared to Baseline - Night-time
Description: as for outcome 8
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 66 | 76 | 72 | 75
Score | -11.5 (32.65) | -6.8 (29.07) | -9.8 (28.73) | -2.2 (28.95)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.006, Mixed model repeated measures; Mean Difference (Final Values) = -11.7, 95% CI 2-sided [-20.0 to -3.3]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.222, Mixed model repeated measures; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-13.0 to 3.0]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.058, Mixed model repeated measures; Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-16.0 to 0.3]

15. Secondary Outcome: Change in the Cough Severity Visual Analogue Scale (VAS) at Week 12 Compared to Baseline - Night-time
Description: as for outcome 8
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 66 | 74 | 68 | 73
Score | -8.9 (35.99) | -7.1 (26.88) | -9.6 (30.24) | -1.5 (33.74)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.027, Mixed model repeated measures; Mean Difference (Final Values) = -10.0, 95% CI 2-sided [-18.9 to -1.2]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.147, Mixed model repeated measures; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-14.9 to 2.2]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.046, Mixed model repeated measures; Mean Difference (Final Values) = -8.9, 95% CI 2-sided [-17.6 to -0.1]

16. Secondary Outcome: Change in the Urge-to-cough Visual Analogue Scale (VAS) at Week 2 Compared to Baseline
Description: The urge-to-cough VAS was a 100 mm scale on which subjects indicated their urge to cough over the previous 24 hours (day/awake time and night time combined). The VAS ranged from "no urge to cough" (0 mm) on the left to "severe urge to cough" (100 mm) on the right. Subjects completed the urge to cough VAS at baseline/Day 1 (pre dose) and at Weeks 2, 4, 8, and 12.
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 72 | 77 | 75 | 74
Score | -20.8 (24.59) | -12.0 (25.09) | -13.8 (22.03) | -7.0 (20.35)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; Change in the urge-to-cough VAS was summarised by treatment group and visit (Weeks 2, 4, 8 and 12) in terms of absolute values and changes from baseline. The effect of treatment in terms of the change from baseline to each scheduled visit (Week 2, Week 4, Week 8 and Week 12) in urge-to cough VAS was analysed using a MMRM with REML estimation; Test type: Superiority; p < 0.001, Mixed model repeated measures; Mean Difference (Final Values) = -12.5, 95% CI 2-sided [-19.5 to -5.5]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.114, Mixed model repeated measures; Mean Difference (Final Values) = -5.5, 95% CI 2-sided [-12.4 to 1.3]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.056, Mixed model repeated measures; Mean Difference (Final Values) = -6.8, 95% CI 2-sided [-13.7 to 0.2]

17. Secondary Outcome: Change in the Urge-to-cough Visual Analogue Scale (VAS) at Week 4 Compared to Baseline
Description: as for outcome 16
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 68 | 77 | 75 | 76
Score | -19.0 (26.93) | -12.0 (26.67) | -17.3 (24.73) | -8.8 (24.26)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.027, Mixed model repeated measures; Mean Difference (Final Values) = -8.9, 95% CI 2-sided [-16.8 to -1.0]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.357, Mixed model repeated measures; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-11.3 to 4.1]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.031, Mixed model repeated measures; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-16.2 to -0.8]

18. Secondary Outcome: Change in the Urge-to-cough Visual Analogue Scale (VAS) at Week 8 Compared to Baseline
Description: as for outcome 16
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 65 | 76 | 72 | 75
Score | -23.8 (28.00) | -14.5 (27.55) | -19.7 (26.80) | -11.0 (24.78)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.008, Mixed model repeated measures; Mean Difference (Final Values) = -11.1, 95% CI 2-sided [-19.2 to -2.9]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.321, Mixed model repeated measures; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-11.8 to 3.9]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.047, Mixed model repeated measures; Mean Difference (Final Values) = -8.1, 95% CI 2-sided [-16.0 to -0.1]

19. Secondary Outcome: Change in the Urge-to-cough Visual Analogue Scale (VAS) at Week 12 Compared to Baseline
Description: as for outcome 16
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 66 | 74 | 68 | 74
Score | -23.7 (27.30) | -12.6 (28.57) | -22.9 (28.43) | -11.8 (26.50)
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.018, Mixed model repeated measures; Mean Difference (Final Values) = -10.1, 95% CI 2-sided [-18.4 to -1.8]
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.682, Mixed model repeated measures; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-9.8 to 6.4]
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.005, Mixed model repeated measures; Mean Difference (Final Values) = -11.8, 95% CI 2-sided [-20.0 to -3.6]

20. Secondary Outcome: Global Rating of Change in Cough Frequency at Week 2
Description: In the Global Rating of Change scale, subjects indicated if there had been a change in their symptoms (cough frequency and, separately, cough severity) since starting the IMP. Subjects responded with "worse", "about the same" or "better". If subjects indicated a change (either "worse" or "better") they then indicated on a 7 point scale the degree of change ranging from 1 (almost the same, hardly any change) to 7 (a very great deal changed). Subjects documented their Global Rating of Change in cough frequency and cough severity at Weeks 2, 4, 8, and 12.
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 73 | 77 | 76 | 74
Participants
  Worse | 4 | 10 | 5 | 11
  About the same | 35 | 37 | 34 | 44
  Better | 34 | 30 | 37 | 19
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; The Global Rating of Change responses were summarised by treatment group and visit (Weeks 2, 4, 8 and 12) as categorical endpoints ("worse", "about the same" and "better"). Pairwise comparisons were performed using the Cochran Mantel Haenszel test stratified by region using modified ridit scores (row mean scores differ); Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.134, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel

21. Secondary Outcome: Global Rating of Change in Cough Frequency at Week 4
Description: as for outcome 20
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 69 | 76 | 74 | 76
Participants
  Worse | 9 | 8 | 6 | 12
  About the same | 32 | 36 | 37 | 39
  Better | 28 | 32 | 31 | 25
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.401, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.175, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.126, Cochran-Mantel-Haenszel

22. Secondary Outcome: Global Rating of Change in Cough Frequency at Week 8
Description: as for outcome 20
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 67 | 75 | 72 | 75
Participants
  Worse | 11 | 17 | 10 | 20
  About the same | 22 | 31 | 37 | 38
  Better | 34 | 27 | 25 | 17
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.144, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.025, Cochran-Mantel-Haenszel

23. Secondary Outcome: Global Rating of Change in Cough Frequency at Week 12
Description: as for outcome 20
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 67 | 74 | 67 | 74
Participants
  Worse | 7 | 13 | 7 | 13
  About the same | 32 | 33 | 31 | 37
  Better | 28 | 28 | 29 | 24
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.158, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.597, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.124, Cochran-Mantel-Haenszel

24. Secondary Outcome: Global Rating of Change in Cough Severity at Week 2
Description: as for outcome 20
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 73 | 77 | 76 | 74
Participants
  Worse | 7 | 8 | 4 | 12
  About the same | 33 | 39 | 35 | 44
  Better | 33 | 30 | 37 | 18
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.01, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.049, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel

25. Secondary Outcome: Global Rating of Change in Cough Severity at Week 4
Description: as for outcome 20
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 69 | 76 | 74 | 76
Participants
  Worse | 9 | 7 | 7 | 14
  About the same | 32 | 43 | 31 | 37
  Better | 28 | 26 | 36 | 25
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.309, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.387, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.025, Cochran-Mantel-Haenszel

26. Secondary Outcome: Global Rating of Change in Cough Severity at Week 8
Description: as for outcome 20
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 67 | 75 | 72 | 75
Participants
  Worse | 8 | 12 | 6 | 15
  About the same | 26 | 36 | 35 | 42
  Better | 33 | 27 | 31 | 18
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.152, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel

27. Secondary Outcome: Global Rating of Change in Cough Severity at Week 12
Description: as for outcome 20
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
Number analyzed (Participants) | 67 | 74 | 67 | 74
Participants
  Worse | 5 | 15 | 8 | 16
  About the same | 38 | 33 | 30 | 36
  Better | 24 | 26 | 29 | 22
Statistical Analysis 1: Comparison: Orvepitant 10mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.100, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Orvepitant 20mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.557, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Orvepitant 30mg vs Placebo; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.054, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Adverse events were reported for each participant from the time of consent up until the last visit (follow-up or early withdrawal). For each completed participant this was a period of 17 weeks.
Description: Adverse events could be volunteered spontaneously by the subject, or were discovered as a result of general, non leading questioning. Note: The adverse events posted in ClinicalTrials.gov results are treatment-emergent adverse events.
Arm/Group | Orvepitant 10mg | Orvepitant 20mg | Orvepitant 30mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/78 | 0/79 | 0/79
Serious Adverse Events (participants affected / at risk) | 1/79 | 1/78 | 3/79 | 1/79
Other Adverse Events (participants affected / at risk) | 63/79 | 48/78 | 53/79 | 40/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orvepitant 10mg (N=79) | Orvepitant 20mg (N=78) | Orvepitant 30mg (N=79) | Placebo (N=79)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orvepitant 10mg (N=79) | Orvepitant 20mg (N=78) | Orvepitant 30mg (N=79) | Placebo (N=79)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (2) | 4 (5) | 3 (3)
Headache (Nervous system disorders) | 7 (7) | 10 (19) | 7 (9) | 4 (6)
Dizziness (Nervous system disorders) | 5 (5) | 4 (4) | 5 (6) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 4 (4) | 5 (5) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 13 (14) | 13 (14) | 11 (11) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 6 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 8 (9) | 7 (10) | 4 (4) | 10 (11)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 4 (5) | 3 (3) | 9 (9)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2) | 3 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT02993822/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT02993822/SAP_002.pdf